CLINICAL TRIAL: NCT00000667
Title: A Phase I/II Dose Escalation Study of Intradermal gp160 to Evaluate Safety, Delayed Type Hypersensitivity (Skin Test) Responses and Immunogenicity in Asymptomatic HIV Seropositive Patients With More Than 400 CD4+ Cells
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Protein Sciences Corporation (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Prevention
Other Study IDs: ACTG 148; 11123 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; Injections, Intradermal; HIV Antigens; HIV Seropositivity; HIV-1; Drug Evaluation; Hypersensitivity, Delayed; AIDS Vaccines; HIV Therapeutic Vaccine
MeSH Terms: conditions — HIV Infections; HIV Seropositivity; Hypersensitivity, Delayed | interventions — VaxSyn HIV-1 (gp160) vaccine

INTERVENTIONS:
Biological: gp160 Vaccine (MicroGeneSys)

SUMMARY:
To determine the safety of intradermal gp160 in HIV seropositive individuals who are asymptomatic and have a relatively intact immune system. To determine whether there is evidence of a delayed-type hypersensitivity (DTH) response (a "positive" skin test) in these patients, and also the dose of gp160 that elicits a delayed-type hypersensitivity (DTH) response. Early immunity to HIV may play an important role in the long interval between virus infection and the onset of clinical disease. Immune responses have been demonstrated in HIV-infected individuals within weeks to months of infection. Although none of these responses has been shown to be protective, it is possible that boosting anti-HIV immune responses through immunization may slow the progression of HIV infection. DTH responses to HIV-derived recombinant envelope glycoprotein could provide a means of measuring an important immune function in infected patients, and serve as an easily measured surrogate marker of cellular immunity. In addition to eliciting local, cutaneous DTH responses, intradermal inoculation of skin test antigens may be immunogenic, resulting in new antibody production and cellular immune responses. This study allows direct comparison of gp160 administered intradermally with alum-adjuvanted intramuscular preparation with respect to immunogenicity in HIV seropositive patients.

DETAILED DESCRIPTION:
Early immunity to HIV may play an important role in the long interval between virus infection and the onset of clinical disease. Immune responses have been demonstrated in HIV-infected individuals within weeks to months of infection. Although none of these responses has been shown to be protective, it is possible that boosting anti-HIV immune responses through immunization may slow the progression of HIV infection. DTH responses to HIV-derived recombinant envelope glycoprotein could provide a means of measuring an important immune function in infected patients, and serve as an easily measured surrogate marker of cellular immunity. In addition to eliciting local, cutaneous DTH responses, intradermal inoculation of skin test antigens may be immunogenic, resulting in new antibody production and cellular immune responses. This study allows direct comparison of gp160 administered intradermally with alum-adjuvanted intramuscular preparation with respect to immunogenicity in HIV seropositive patients.

Each of 10 volunteers is initially injected with the lowest dose of intradermal antigen and the injection site observed at 24, 48, and 72 hours. Clinical and laboratory evaluations are performed 4 and 8 weeks after inoculation. If there is not delayed-type hypersensitivity (DTH) response to the lowest dose, patients are retested at the next dose 8 weeks later and dose escalation is continued at 8-week intervals until (1) there is a DTH response to gp160; or (2) the maximum anticipated dose is reached. In any individual, a higher dosage is administered only if there is no evidence of DTH response. Patients with a DTH may continue to receive booster injections of gp160 at 3 month intervals up to week 70. Patients with an immune response but no DTH may continue to receive injections for an additional year. A second group of 10 asymptomatic individuals are recruited and inoculated with the dose found to bring about either a DTH or lymphocyte proliferative response in 7 of the 10 patients in the first group. If the second group confirms the results of the initial group, the study is amended to include patients with AIDS-related complex (ARC) and AIDS.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Acute use (< 14 days) of acyclovir for Herpes simplex virus infections or ketoconazole for symptomatic Candida infections.

Patients must have the following:

* Asymptomatic HIV seropositivity.
* Patients with CD4 counts of 400 - 500 cells/mm3 must be informed of the recommended zidovudine (AZT) therapy and sign an informed consent statement declining AZT therapy.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Systemic symptoms other than lymphadenopathy thought to be due to HIV infection including:
* Fatigue/malaise of > 1 month duration that interferes with normal activities.
* Fever of > 100 degrees F persisting for > 15 in a 30-day interval without definable cause.
* Involuntary weight loss in excess of 10 pounds or > 10 percent of normal weight within a 6-month interval.
* Diarrhea (> 3 stools/day) persisting for more than 30 days without definable cause.
* Recurrent oral candidiasis.
* Multidermatomal herpes zoster.
* Biopsy proven hairy leukoplakia.
* Evidence of clinically significant central nervous system dysfunction as assessed by neurological exam.

Concurrent Medication:

Excluded:

* Antiretroviral agents of proven or potential efficacy.
* Any potential immunoenhancing or immunosuppressive drugs.

Patients with the following are excluded:

* Known hypersensitivity to insect cells or baculovirus.
* Abnormal chest x-ray taken within 3 months of study entry.
* Systemic symptoms other than lymphadenopathy thought to be due to HIV infection as listed in the patient exclusion coexisting diseases or complications.
* Evidence of clinically significant central nervous system dysfunction as assessed by neurological exam.
* Unwilling or unable to give written informed consent.

Prior Medication:

Excluded within 90 days of study entry:

* Zidovudine (AZT).
* Didanosine (ddI).
* Any potential antiretroviral.
* Immunomodulating agents.

Active substance abuse (either continuing daily alcohol abuse or intravenous drug use).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Study Completion 1993-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katzenstein DA, Study Chair
Locations (1):
- NY Univ. HIV/AIDS CRS, New York, New York, United States

REFERENCES:
- [Background] Katzenstein D, Valentine F, Kundu S, Haslett P, Smith G, Merigan T. Delayed-type-hypersensitivity reactions to intradermal gp160 in HIV infected individuals immunized with gp160. Int Conf AIDS. 1992 Jul 19-24;8(2):A35 (abstract no PoA 2192)
- [Background] Katzenstein DA, Kundu S, Spritzler J, Smoller BR, Haszlett P, Valentine F, Merigan TC. Delayed-type hypersensitivity to recombinant HIV envelope glycoprotein (rgp160) after immunization with homologous antigen. J Acquir Immune Defic Syndr. 1999 Dec 1;22(4):341-7. doi: 10.1097/00126334-199912010-00004. PMID 10634195